CLINICAL TRIAL: NCT01043991
Title: Intracoronary Injection of Epo During Reperfusion in Patients Hospitalized for First Acute Myocardial Infarct STEMI
Brief Title: Intracoronary Injection of Epo After Myocardial Infarct "Intra-CO-EpoMI"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8042
Record Dates: First submitted 2009-09-22; First posted 2010-01-07 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Acute Myocardial Infarct
Keywords: STEMI; AMI,; acute myocardial infarct; Epo; Erythropoietin; ischemia-reperfusion; apoptosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO (Experimental): single bolus of EPO, 150 µg
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator): NaCl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa
  Arms: EPO
Drug: Placebo
  Arms: Placebo

SUMMARY:
Primary endpoint: Is intracoronary injection of a single dose of darbepoetin alpha, during reperfusion in patients hospitalized for ST segment elevation myocardial infarction (STEMI), able to reduce infarct size ?

In in vivo studies, many experiments evidenced infarct size reduction, due to anti-apoptotic compounds, when given during reperfusion, after cardiac ischemia. In humans, post-conditioning offers such a protection, as the investigators have previously showed (Staat P et al. Post-conditioning the human heart. Circulation. 2005 112(14):2143-8).

Infarct size reduction could lead to a reduced rate of complications (heart failure, rhythmic complications) and finally, morbidity and even mortality. This protection depends on anti-apoptotic properties (Zhao ZQ et al. Inhibition of myocardial injury by ischemic postconditioning during reperfusion: comparison with ischemic preconditioning. Am J Physiology Heart Circ Physiology 2003 Aug; 285(2):H579-88). Many drugs have been proposed to be able to mimic this phenomenon. Among them, many are efficient but toxic in vivo or difficult to manage (insulin, morphin). One of the most promising agent could then be erythropoietin (EPO) (Opie LH et al. Postconditioning for protection of the infarcting heart. Lancet. 2006; 367(9509):456-8). In order to target ischemia-reperfusion injuries, EPO impact is better and better demonstrated (e.g.: Mudalagiri NR. Erythropoietin protects the human myocardium against hypoxia and reoxygenation injury via phosphatidylinositol-3 kinase and ERK1-2 activation. Br J Pharmacol. 2007 Oct 22). The purpose of the study is to test this hypothesis in humans, on the onset of the reperfusion, after myocardial ischemia (acute myocardial infarct). EPO could contribute to protect myocardium against ischemia-reperfusion injury. This impact could rely on anti-apoptotic properties.

DETAILED DESCRIPTION:
Multiple Centers.:

5 centers located in France:

* Montpellier
* Clermont-Ferrand
* Lyon
* Marseille
* Nîmes

Study design: Open-label, placebo-controlled, single-blinded. Patient in treatment group will receive intracoronary single bolus of EPO (150 µg), as soon as significant reperfusion is obtained (as measured by TIMI flow 2 or 3). In control group, placebo will be used. Placebo must be presented exactly the same as the drug.

Length of Treatment: One shot during reperfusion procedure.

Follow-up Period: 72nd hour post-admission for plasma kinetics of cardiac enzymes 5th to 7th day after revascularization procedure for MRI measurements, and echocardiography3th month post-MI MRI, echocardiography3th month: phone contact.

Sample Size: 27 patients in each arm, 54 patients total.

ELIGIBILITY:
Inclusion Criteria:

* ACS with persistent ST elevation
* First episode
* Symptoms onset < 12 hours
* Eligible for angioplasty
* Culprit coronary artery occluded (TIMI flow 0-1) at admission, and then adequately reperfused (TIMI flow 2-3) prior to EPO injection

Exclusion Criteria:

* Cardiogenic shock
* Cardiac arrest
* Currently receiving EPO
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging (MRI) determination of infarct size | 12 weeks

SECONDARY OUTCOMES:
Cardiac enzymes | 12 weeks
Echocardiography | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PIOT, Pr, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

REFERENCES:
- [Derived] Roubille F, Micheau A, Combes S, Thibaut S, Souteyrand G, Cayla G, Bonello L, Lesavre N, Sportouch-Dukhan C, Klein F, Berboucha S, Cade S, Cung TT, Raczka F, Macia JC, Gervasoni R, Cransac F, Leclercq F, Barrere-Lemaire S, Paganelli F, Mottref P, Vernhet Kovacsik H, Ovize M, Piot C. Intracoronary administration of darbepoetin-alpha at onset of reperfusion in acute myocardial infarction: results of the randomized Intra-Co-EpoMI trial. Arch Cardiovasc Dis. 2013 Mar;106(3):135-45. doi: 10.1016/j.acvd.2012.12.001. Epub 2013 Feb 1. PMID 23582675